CLINICAL TRIAL: NCT02836639
Title: Phase II Study for Safety and Efficacy of BEB (Bendamustine, Etoposide, Busulfan) Conditioning Regimen for ASCT in Non-Hodgkin's Lymphoma
Brief Title: BEB Conditioning Regimen for Autologous Stem-cell Transplantation(ASCT) in Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Ho-Jin Shin, Professor department of hematooncology, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEB
Record Dates: First submitted 2016-06-27; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Busulfan; Etoposide; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan, Etoposide, Bendamustine (Experimental): All patients will receive the conditioning regimen followed by autologous stem cell transplantation.
  Interventions: Drug: Busulfan; Drug: Etoposide; Drug: Bendamustine

INTERVENTIONS:
Drug: Busulfan — Busulfan 0.8 mg/kg four times per day from day -7 to day -5
Drug: Etoposide — Etoposide 400 mg/m2 from day -5 to day -4
Drug: Bendamustine — Bendamustine 200 mg/m2 starting dose on day -3 and -2

SUMMARY:
Phase II study for safety and efficacy of BEB (Bendamustine, Etoposide, Busulfan) conditioning regimen for ASCT in non-Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically diagnosed non-Hodgkin's lymphoma
2. 16 ≤ Age ≤ 65 years
3. Adequate cardiac function with cardiac ejection fraction greater than 50% by echocardiogram or multiple gated acquisition scan(MUGA)
4. Adequate kidney function with serum creatinine< 2.0 mg/dL
5. Adequate liver function with /serum bilirubin lower than 2 times the normal upper limit, Aspartate aminotransferase(AST)/ Alanine aminotransaminase(ALT) lower than 3 times the normal upper limit. In case of DLBCL liver invasion; serum bilirubin lower than 5 times the normal upper limit, AST/ALT lower than 5 times the normal upper limit.
6. Adequate bone marrow function with absolute neutrophil count ≥ 1,500/µL; platelets ≥ 75,000/µL; hemoglobin ≥ 9.0 g/dL
7. Patients who voluntarily gave informed consent before performing any test that is not part of routine care of patients
8. Candidate for ASCT

Exclusion Criteria:

1. Positive serology for HIV, hepatitis C virus(HCV) If the hepatitis B virus(HBV) patient was administrated prophylactic antiviral agents. It would be eligible following the judgment of the investigator
2. Pregnant or breast-feeding. Females of childbearing potential who do not agree to undergo pregnancy tests or repeated use effective birth control while included in the clinical trial.
3. Patients with serious or uncontrolled medical condition; 1) Abnormalities in cardiac function or clinically significant heart disease such as congestive heart failure, arrhythmia, unstable angina with treatment within 6 months or acute myocardial infarction; 2) Previous history of serious neurological or psychiatric disease; 3) Acute, severe active infection requiring immediate treatment(Virus, Bacteria, Fungal infection); 4) chronic obstructive pulmonary disease requiring oral steroid therapy or Forced expiratory volume 1 sec(FEV1)<0.8 L less than the test of pulmonary function at rest; 5) If there are other diseases that are deemed inappropriate as a target of the present clinical trial following the Investigator's judgment; 6) Congenital or acquired bleeding disorders
4. Patients receiving any other investigational systemic therapy (Hormone, Immune, chemotherapy)
5. Allergic to the investigational drug
6. Patients who have difficulty understanding the informed consent form or patients who did not give consent
7. Serum bilirubin upper than 2 times the normal upper limit
8. Major surgery procedure within 30 days prior to start of investigational treatment
9. Patients vaccinated against yellow fever

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year after ASCT
Progression-free survival | 3 years after ASCT

SECONDARY OUTCOMES:
Overall survival | 1 year and 3 year after ASCT
Complete response rate | 1 year and 3 year after ASCT
Incidence of adverse events | 1 year and 3 year after ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Shin, Principal Investigator — Pusan National Universty Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visani G, Malerba L, Stefani PM, Capria S, Galieni P, Gaudio F, Specchia G, Meloni G, Gherlinzoni F, Giardini C, Falcioni S, Cuberli F, Gobbi M, Sarina B, Santoro A, Ferrara F, Rocchi M, Ocio EM, Caballero MD, Isidori A. BeEAM (bendamustine, etoposide, cytarabine, melphalan) before autologous stem cell transplantation is safe and effective for resistant/relapsed lymphoma patients. Blood. 2011 Sep 22;118(12):3419-25. doi: 10.1182/blood-2011-04-351924. Epub 2011 Aug 3. PMID 21816830
- [Background] Shin HJ, Lee WS, Lee HS, Kim H, Lee GW, Song MK, Kim JS, Yhim HY, Chung JS. Busulfan-containing conditioning regimens are optimal preparative regimens for autologous stem cell transplant in patients with diffuse large B-cell lymphoma. Leuk Lymphoma. 2014 Nov;55(11):2490-6. doi: 10.3109/10428194.2014.882504. Epub 2014 Mar 7. PMID 24432893